CLINICAL TRIAL: NCT03460288
Title: Computer-based Training (Retraining) for People With Gambling Problems
Acronym: Retraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Retraining
Record Dates: First submitted 2018-02-05; First posted 2018-03-09 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Gambling, Pathological
Keywords: Gambling, Problematic Gambling, Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: The study is a randomly controlled study with 2 conditions: Condition 1: Computer-based training program (retraining), condition 2: Wait-list control group (access to the training after the post-assessment).
  Two assessments-points, the intervention period (pre-post) is eight weeks. Sociodemographic and pathological data are obtained with an internet survey on Unipark®.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The training-program includes ten pictures related to slot-machine gambling and 10 neutral pictures that need to be either pushed (i.e., avoidance) or pulled (i.e., approach) with the computer mouse or finger (when a tablet is used) according to a non-affective dimension (color of the frame). Pictures are presented in random order.
  Interventions: Behavioral: Retraining (AAT)
- Wait-list control group (No Intervention): The participants of the wait-list control condition do not receive the retraining intervention during the intervention period of 8 weeks, but may continue any treatment that has already been started before, including pharmacological treatment. Participants in the wait-list control condition receive full access to the training program after completion of the post-assessment.

INTERVENTIONS:
Behavioral: Retraining (AAT) — The training program is based upon the approach-avoidance task (AAT) and can be easily performed on a computer, laptop or tablet. There is a total of 20 pictures, 10 slot-machine gambling related pictures and 10 neutral pictures that were already used in a prior study (Wittekind et al., submitted). The pictures appear on the computer screen and have to be either pushed or pulled. Pushing and pulling depends on a masked instruction (not related to the content of the pictures, but to the color of the frame). All gambling-related pictures are framed with the color that is instructed to be pushed, all neutral pictures are framed with the color that is instructed to be pulled.
  Arms: Intervention Group

SUMMARY:
The study examines the efficacy and acceptance of a computer-based training program for individuals with problematic or pathological gambling behavior. The study intends to investigate the extent to which the computer-based training program leads to a significant reduction in pathological gambling (primary outcome) when compared to a control group. The study design is a randomized-controlled trial with one intervention group and one wait-list control group.

DETAILED DESCRIPTION:
The study examines the efficacy of a computer-based training program for individuals with problematic and pathological gambling behavior. The main objective of the study is to investigate the extent to which the online program leads to a significant reduction in pathological gambling. The primary outcome is the Pathological Gambling Adaptation of the Yale-Brown Obsessive Compulsory Scale (PG-YBOCS total score) as a measure of the severity of pathological gambling symptoms. Secondary outcomes are further measures of gambling-related symptoms, such as the South Oaks Gambling Screen (SOGS), as well as rates of depression, measured with the Patient Health Questionnaire - 9 items depression module (PHQ-9), and rates of impulsivity, measured with the impulsivity subscale of the Eysenck's Impulsivity Inventory (I-7). The training is expected to lead to a significant reduction in problematic/pathological gambling behavior (PG-YBOCS) and all secondary outcomes when compared to a control group. The study design is a randomized-controlled trial with one intervention group and one wait-list control group and two assessment times (pre and post). The intervention group receives the download link for the training program directly following the baseline survey and can use the training over a period of 8 weeks, whereas the wait-list control group receives access to the training after completion of the post-survey.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* access to internet
* sufficient command of the German language
* willingness to participate in two short (25-30 minutes) online surveys
* willingness to use the online program over a period of 8 weeks (participants who do not use the program are also included in the analysis)
* willingness to leave an (anonymous) email-address
* subjective need for treatment

Exclusion Criteria:

* presence of a lifetime diagnosis of schizophrenia or bipolar disorder
* acute suicidal tendency (assessed with item 9 of the PHQ-9, ≥3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Pathological Gambling Adaptation of Yale-Brown Obsessive Compulsive Scale (PG-YBOCS) | Change in PG-YBOCS from pre- to post-intervention (i.e. 8 week interval)
  The total score consists of ten items that measure the severity of gambling symptoms within the past week. The first five questions assess urges and thoughts associated with gambling, whereas the last five questions assess the behavioral component of the disorder. The sum score of each subscale ranges from 0-20. Each subscale can be analyzed separately as well as together as a total score (primary outcome). The total score can be interpreted as follows: 0-7: sub-clinical, 8-15: mild, 16-23: moderate, 24-31: severe and 32-40: extreme gambling symptoms.

SECONDARY OUTCOMES:
South Oaks Gambling Screen (SOGS) | Change in SOGS from pre- to post-intervention (i.e. 8 week interval)
  20-items self-report measure to screen for engagement in gambling activities and gambling-related problems. A score between 0-2 corresponds to non-problematic gambling, a score of 3-4 to at-risk gambling, and a score of 5-20 to probable pathological gambling.
Eysenck Impulsiveness Questionnaire - Subscale Impulsivity (I-7) | Change in I-7 from pre- to post-intervention (i.e. 8 week interval)
  Impulsivity will be assessed with the 17-item impulsivity subscale of the Eysenck Impulsiveness Questionnaire, which consists of the three subscales impulsiveness, venturesomeness, and empathy (Eysenck, Pearson, Easting, & Allsopp, 1985). The reliability of the subscale is good (α = .82 - .85).
Patient Health Questionnaire - 9 items depression module (PHQ-9) | Change in PHQ-9 from pre- to post-intervention (i.e. 8 week interval)
  The PHQ-9 is used to assess depressive symptoms over the past week. The nine items of the questionnaire are based upon the diagnostic criteria of major depression. Internal consistency of the scale is very good (Cronbach´s α = .86 - .89).

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany